CLINICAL TRIAL: NCT04277611
Title: Comparison Between Ultrasound Guided Subcostal Oblique Quadratus Lumborum Block and Erector Spinae Plane Block in Patients Undergoing Percutaneous Nephrolithotomy
Brief Title: Comaprison Between QLB and ESPB in Patients for PCNL Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Peter Bassem Halim Gadelsyed, Resident Doctor in Anesthesia, postoperative ICU and pain management department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: QLB and ESPB comparison
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Pain, Postoperative
Keywords: pain management; Nephrolithotomy; QLB; ESPB; Erector Spinae; Quadratus Lumborum; Anesthesia; ultrasound; regional anethesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QLB (Active Comparator): The patient is in the prone position, an ultrasound probe is placed in a transverse, oblique, and paramedian orientation approximately lateral to the posterior axillary line. The needle is then inserted in-plane from the medial side of the transducer and advanced laterally to enter the interfascial plane between the Quadratus Lumborum muscle and the kidney. We confirmed that the local anesthetic appeared to press down the kidney in the ultrasound image
  Interventions: Procedure: Subcostal Oblique Quadratus Lumborum Block and Erector Spinae Plain Block.
- ESPB (Active Comparator): Using aseptic technique, an ultrasound probe is placed at the T9 vertebral level. After identifying the ribs and sliding towards the midline in a longitudinal parasagittal orientation, the overlying Erector Spinae is identified by visualization of the transition between the rib and transverse apophysis a block needle is inserted in plane with ultrasound beam and is advanced in a cephalo-caudal direction until the tip contacted the transverse process.
  Interventions: Procedure: Subcostal Oblique Quadratus Lumborum Block and Erector Spinae Plain Block.

INTERVENTIONS:
Procedure: Subcostal Oblique Quadratus Lumborum Block and Erector Spinae Plain Block. — patients undergo general anesthesia,will be put in prone position.In case of Quadratus Lumborum block 1-3 mL of normal saline is injected to produce hydro-dissection and spread cranially between the QL and kidney. The corresponding ultrasonographic sign is a lunar-shaped hypo-echoic fluid collection observed between the long axis of the kidney and QL muscle. 20 ml Bupivacaine 0.5%, 10 ml Lidocaine 2%, and 10 ml normal saline is administered. In case of the ESPB The location of the needle tip is confirmed by hydro-dissection and after visualizing the fluid spread lifting the Erector Spinae off the transverse process, 20 ml bupivacaine 0.5%, 10 ml Lidocaine 2%, and 10 ml normal saline is injected.

SUMMARY:
comparing the subcostal oblique Quadratus Lumborum block and the Erector Spinae plane block in patients undergoing percutaneous nephrolithotomy operation to get the best and longest postoperative analgesic effect.

DETAILED DESCRIPTION:
Here the investigators are going to compare between the Anterior approach for the subcostal oblique Quadratus Lumborum block (QLB) and the Erector Spinae Plane Block (ESPB) to determine their level of spread and their value in controlling postoperative pain in patients scheduled for Percutaneous Nephrolithotomy surgery. We hypothesized that quadratus lumborum is not inferior regarding the duration of analgesia when compared to erector spinae in patients undergoing percutaneous nephrolithotomy under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Both sex
* Age: 18-60
* ASA (American Society of Anesthesiologists) class I and II
* Elective surgery
* Patients undergoing PNL surgery

Exclusion Criteria:

* Patient's refusal
* Allergy or contraindications to drugs used in the study
* Emergency surgery
* Psychiatric disorders
* Severely co-morbid patients
* Inflammation or infection over injection site
* Bleeding diathesis; INR more than 1.5 and Platelet count less than 100,000/mm3
* Peripheral neuropathy
* Obese patients BMI ≥35
* Patients on previous opioid therapy
* Pre-operative haemoglobin <10 mg/dl
* Inability to properly describe postoperative pain to investigators
* Coagulation abnormalities
* History of drug addiction or alcohol abuse
* History of Previous renal surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Analgesia | 48 hours
  Total opioid consumption during the first 48hours postoperatively.

SECONDARY OUTCOMES:
Analgesia | 24 hours
  first Analgesic request postoperatively.
episodes of nausea and vomiting | within 24 hours postoperative
  to investigate if there is or not.
Pain Scores using Visual Analog Scale (VAS) Scores | 24 hours postoperative.
  VAS is a scale to determine the patient's pain level.
ambulation time | 5 days postoperative
  time from the end of the surgery to the first time to out-of-bed activity
time of recovery of bowl movement | 5 days postoperative
  time from the end of the surgery to the first time of bowl movement
patient satisfaction with anesthesia | 48 hours postoperative.
  Patient satisfaction with anesthesia was assessed using a 5-point scale (5: very satisfied; 4: satisfied; 3: neither satisfied nor dissatisfied; 2: dissatisfied; 1: very dissatisfied)
postoperative length of hospital stay | within 2 weeks postoperative.
  till time of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Amr Thabet, Lecturer, Study Director — Assiut University; Alaa Attia, Professor, Study Chair — Assiut University
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No